CLINICAL TRIAL: NCT01029197
Title: Multicomponent Cognitive Behavioral Therapy for Posttraumatic Stress Disorder and Substance Abuse: A Pilot Study
Brief Title: Multicomponent Cognitive Behavioral Therapy(CBT) for Posttraumatic Stress Disorder (PTSD) and Substance Abuse
Acronym: PTSD/SUD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Karen Cusack, Ph.D., University of North Carolina at Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5K01MH079343 (NIH)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Posttraumatic Stress Disorder; Substance Abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Implosive Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT Intervention (Experimental): The CBT intervention includes psychoeducation and coping and social skills delivered in a group format, and exposure therapy delivered in individual sessions
  Interventions: Behavioral: CBT and exposure therapy for PTSD
- Treatment as Usual (Active Comparator): The TAU Condition will receive usual services at the community clinic, which may include medications, individual or group therapy
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: CBT and exposure therapy for PTSD — The CBT intervention will be administered twice weekly in group therapy sessions for 7 weeks, and then twice weekly individual sessions for 4 weeks.
  Arms: CBT Intervention
Other: Treatment as Usual — Participants in the treatment as usual condition will receive their usual services at the community clinic where they receive mental health and substance abuse services
  Arms: Treatment as Usual

SUMMARY:
Purpose: To conduct a pilot study of a cognitive-behavioral treatment (CBT) for PTSD and substance abuse among persons with serious mental illness (SMI) treated in a community setting.

Participants: Participants will be 50 volunteer adult individuals with PTSD and substance use disorders (SUD), and SMI who are receiving services at the Freedom House Recovery Center, served through the Orange Person Chatham (OPC) Area Program.

Procedures (methods): Participants will be randomly assigned to one of two conditions: 1) the CBT intervention plus treatment as usual; or, 2) treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Currently receiving services at Freedom House
* Meet DSM-IV criteria for PTSD
* Meet criteria for Substance Use Disorder
* Able to understand and provide informed consent

Exclusion Criteria:

• Psychiatric hospitalization or suicide attempt in the past two months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale | 3 months

SECONDARY OUTCOMES:
Addiction Severity Index | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Cusack, PhD, Principal Investigator — University of North Carolina, Chapel Hill; William Blair, B.S., Study Director — University of North Carolina, Chapel Hill
Locations (1):
- Freedom House, Chapel Hill, North Carolina, United States